CLINICAL TRIAL: NCT05215444
Title: Evaluation of Some Prognostic Factors in Acute Aluminum Phosphide Intoxicated Cases
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, shymaa mohamed nasrallah abdulrhman, demonstrator, Zagazig University
Other Study IDs: 6665
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Aluminum Phosphide Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 cm of blood will be collected from included patients on admission, 2cm in tube contain EDTA to perform CBC test and 8 cm will be transferred to a dry clean centrifuge tube and will be left upright to clot then it will be centrifuged for 10 minutes at 5000rpm, the serum will be separated and preserved at -80°C to be used later for further biochemical analyses
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- survivors
  Interventions: Diagnostic Test: some prognostic factors
- non survivors
  Interventions: Diagnostic Test: some prognostic factors

INTERVENTIONS:
Diagnostic Test: some prognostic factors — cortisol level, renin, troponin I, MDA ,catalase, super oxide dismutase, liver functions, kidney functions, arterial blood gases, sodium level, potassium level. white blood cells count

SUMMARY:
study of some laboratory and clinical findings which may show the severity of aluminium phosphide toxicity and the need of the cases to be admitted to ICU

DETAILED DESCRIPTION:
aluminium phosphide poisoning is a major cause of death in intoxicated and suicidal cases since there is no antidote and there is no specific investigation for it so there is a need for further study to identify the cause of death and the most specific investigation in the case of AlP toxicity

ELIGIBILITY:
Inclusion Criteria:

1. History of exposure or intake of Aluminum phosphide.
2. Clinical picture of Acute Aluminum phosphide poisoning including severe vomiting, hypotension, abdominal pain, cardio-pulmonary distress.
3. Cases of the age of 15 to 45 years old

Exclusion Criteria:

- 1. Cases with an unclear history. 2. History of co-morbidities or systemic diseases because of the possibility of misleading laboratory results.

3. History of co-ingestion of drugs or another poison.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: the mode of toxicity is suicidal by ingestion of AlP tablet
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
prognosis | the first 24 post poisoning
  predict the mortality of intoxicated AlP cases

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No